CLINICAL TRIAL: NCT02552121
Title: Dose-escalating and Cohort Expansion Safety Trial of Tissue Factor Specific Antibody Drug Conjugate Tisotumab Vedotin (HuMax®-TF-ADC) in Patients With Locally Advanced and/or Metastatic Solid Tumors Known to Express Tissue Factor
Brief Title: Tisotumab Vedotin (HuMax®-TF-ADC) Safety Study in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GEN702; innovaTV 202 (Other: Genmab)
Record Dates: First submitted 2015-09-14; First posted 2015-09-16 (Estimated); Results first posted 2019-03-12 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Ovary Cancer; Cervix Cancer; Endometrium Cancer; Bladder Cancer; Prostate Cancer (CRPC); Esophagus Cancer; Lung Cancer (NSCLC)
Keywords: ovary cancer; cervix cancer; endometrium cancer; bladder cancer; prostate cancer (CRPC); esophagus cancer; lung cancer (NSCLC)
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Urinary Bladder Neoplasms; Prostatic Neoplasms; Esophageal Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — tisotumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Tisotumab vedotin (HuMax-TF-ADC) (Experimental)
  Interventions: Drug: Tisotumab vedotin (HuMax-TF-ADC)

INTERVENTIONS:
Drug: Tisotumab vedotin (HuMax-TF-ADC)

SUMMARY:
The purpose of the trial is to establish the tolerability of tisotumab vedotin (HuMax-TF-ADC) dosed three times every four weeks (3q4wk) in a mixed population of patients with specified solid tumors.

DETAILED DESCRIPTION:
The study is conducted in two parts. In the Dose Escalation portion of the trial, subjects are enrolled into cohorts at increasing dose levels of tisotumab vedotin (HuMax-TF-ADC) in 28 day treatment cycles.

The Cohort Expansion portion of the trial will further explore the recommended phase 2 dose of tisotumab vedotin (HuMax-TF-ADC) as determined in Part 1.

ELIGIBILITY:
Inclusion Criteria:

- Patients with relapsed, advanced and/or metastatic cancer who have failed available standard treatments or who are not candidates for standard therapy.

Patients must have measurable disease according to RECIST v1.1

* Age ≥ 18 years.
* Acceptable renal function.
* Acceptable liver function.
* Acceptable hematological status (hematologic support allowed under certain circumstances).
* Acceptable coagulation status.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of at least three months.
* A negative serum pregnancy test (if female and aged between 18-55 years old).
* Women who are pregnant or breast feeding are not to be included.
* Patients, both females and males, of reproductive potential must agree to use adequate contraception during and for six months after the last infusion of HuMax-TF-ADC.
* Following receipt of verbal and written information about the study, patients must provide signed informed consent before any study-related activity is carried out.

Exclusion Criteria:

* Known past or current coagulation defects.
* Diffuse alveolar hemorrhage from vasculitis.
* Known bleeding diathesis.
* Ongoing major bleeding.
* Trauma with increased risk of life-threatening bleeding.
* Have clinically significant cardiac disease.
* A baseline QT interval as corrected by Fridericia's formula (QTcF) > 450 msec, a complete left bundle branch block (defined as a QRS interval ≥ 120 msec in left bundle branch block form) or an incomplete left bundle branch block.
* Therapeutic anti-coagulative or long term anti-platelet treatment except use of low dose acetylsalicylic acid (ASA) up to 81 mg/day and non-ASA nonsteroidal anti-inflammatory drugs (NSAIDs).
* Have received granulocyte colony stimulating factor (G-CSF) or granulocyte/macrophage colony stimulating factor support within one week or pegylated G-CSF within two weeks before the Screening Visit.
* Have received a cumulative dose of corticosteroid ≥ 150 mg (prednisone or equivalent doses of corticosteroids) within two weeks before the first infusion.
* No dietary supplements allowed during the study period, except multivitamins, vitamin D and calcium.
* Major surgery within six weeks or open biopsy within 14 days before drug infusion.
* Plan for any major surgery during treatment period.
* Patients not willing or able to have a pre-trial tumor biopsy taken (the screening biopsy can be omitted if archived material is available).
* Presence or anticipated requirement of epidural catheter in relation to infusions (within 48 hours before and after dose of trial drug).
* Any history of intracerebral arteriovenous malformation, cerebral aneurysm, brain metastases or stroke.
* Any anticancer therapy including; small molecules, immunotherapy, chemotherapy monoclonal antibodies or any other experimental drug within four weeks or five half lives, whichever is longest, before first infusion.
* Prior treatment with bevacizumab within twelve weeks before the first infusion.
* Prior therapy with a conjugated or unconjugated auristatin derivative.
* Radiotherapy within 28 days prior to first dose.
* Patients who have not recovered from symptomatic side effects of radiotherapy at the time of initiation of screening procedure.
* Known past or current malignancy other than inclusion diagnosis, except for:
* Cervical carcinoma of Stage 1B or less.
* Non-invasive basal cell or squamous cell skin carcinoma.
* Non-invasive, superficial bladder cancer.
* Prostate cancer with a current PSA level < 0.1 ng/mL.
* Breast cancer in BRCA1 or BRACA2 positive ovarian cancer patients.
* Any curable cancer with a complete response (CR) of > 5 years duration.
* Radiographic evidence of cavitating pulmonary lesions and tumor adjacent to or invading any large blood vessel unless approved by sponsor.
* Ongoing, significant , uncontrolled medical condition.
* Presence of peripheral neuropathy.
* Active viral, bacterial or fungal infection requiring intravenous treatment with antimicrobial therapy starting less than four weeks prior to first dose.
* Oral treatment with antimicrobial therapy starting less than two weeks prior to first dose.
* Known human immunodeficiency virus seropositivity.
* Positive serology (unless due to vaccination or passive immunization due to Ig therapy) for hepatitis B.
* Positive serology for hepatitis C based on test at screening.
* Inflammatory bowel disease including Crohn's disease and colitis ulcerosa.
* Inflammatory lung disease including moderate and severe asthma and chronic obstructive pulmonary disease (COPD) requiring chronic medical therapy.
* Ongoing acute or chronic inflammatory skin disease.
* Active ocular surface disease at baseline (based on ophthalmological evaluation).
* History of cicatricial conjunctivitis (as evaluated by an ophthalmologist).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johann de Bono, Professor, Principal Investigator — The Institute of Cancer Research & The Royal Marsden NHS Foundation Trust
Locations (16):
- MD Anderson Cancer Center, Houston, Texas, United States
- Belgium (7):
  - Institut Jules Bordet, Brussels, Brussels Capital
  - Universitaire Ziekenhuizen Leuven, Leuven, Flemish Brabant
  - Grand Hôpital de Charleroi, Charleroi, Hainaut
  - CHU de Liège, Liège, Liège
  - CHU UCL Namur - site Godinne, Yvoir, Namur
  - Cliniques Universitaires Saint-Luc, Brussels
  - CHU UCL Namur - Sainte Elisabeth, Namur
- Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark
- Hungary (3):
  - Petz Aladár Megyei Oktató Kórház, Győr, Győr-Moson-Sopron
  - Debreceni Egyetem Klinikai Központ, Debrecen, Hajdú-Bihar
  - Semmelweis Egyetem Onkológiai Központ, Budapest
- United Kingdom (4):
  - University College London Hospitals NHS Foundation Trust, London, England
  - Sarah Cannon Cancer Center, London, England
  - The Christie NHS Foundation Trust, Manchester, England
  - The Royal Marsden NHS Foundation Trust, Sutton

REFERENCES:
- [Derived] Feng S, Gunawan R, Passey C, Voellinger J, Polhamus D, Gerritsen A, O'Day C, Carret AS, Soumaoro I, Gupta M, Hanley WD. Exposure-safety Markov modeling of ocular adverse events in patient populations treated with tisotumab vedotin. J Pharmacokinet Pharmacodyn. 2025 Oct 3;52(5):55. doi: 10.1007/s10928-025-10003-w. PMID 41044356
- [Derived] Passey C, Voellinger J, Gibiansky L, Gunawan R, Nicacio L, Soumaoro I, Hanley WD, Winter H, Gupta M. Exposure-safety and exposure-efficacy analyses for tisotumab vedotin for patients with locally advanced or metastatic solid tumors. CPT Pharmacometrics Syst Pharmacol. 2023 Sep;12(9):1262-1273. doi: 10.1002/psp4.13007. Epub 2023 Jul 26. PMID 37496366

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For the Dose Escalation, participants took part in the trial at 3 sites located in Denmark, the United Kingdom (UK), and the United States (USA) from 30 Nov 2015 until 10 Feb 2017. Cohort Expansion trial was performed at 10 sites located in Belgium, UK, Denmark, and the USA from 16 Feb 2016 until the last participant visit on 13 Dec 2017.
Groups:
- Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg: Tisotumab vedotin 0.9 mg/kg was administered as an intravenous infusion, over a minimum of 30 minutes, 3 times every 4 weeks (3q4wk).
- Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg: Tisotumab vedotin 1.2 mg/kg was administered as an intravenous infusion, over a minimum of 30 minutes, 3 times every 4 weeks (3q4wk).
- Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian: Participants with the indication of ovarian cancer, received Tisotumab vedotin 1.2 mg/kg (the recommended dose for phase II trials [RP2D] from the Dose Escalation part), administered as an intravenous infusion, over a minimum of 30 minutes 3 times every 4 weeks (3q4wk).
- Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical: Participants with the indication of cervical cancer, received Tisotumab vedotin 1.2 mg/kg (the recommended dose for phase II trials [RP2D] from the Dose Escalation part), administered as an intravenous infusion, over a minimum of 30 minutes 3 times every 4 weeks (3q4wk).
- Part 2 Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian: Participants with the indication of ovarian cancer, received Tisotumab vedotin 1.2 mg/kg (RP2D from the Dose Escalation part), administered as an intravenous infusion, over a minimum of 30 minutes 3 times every 4 weeks (3q4wk). Due to severe ocular toxicity, participants switched to receive Tisotumab vedotin at 2.0 mg/kg, administered as an intravenous infusion once every 3 weeks (1q3w).
- Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical: Participants with the indication of cervical cancer, received Tisotumab vedotin 1.2 mg/kg (RP2D from the Dose Escalation part), administered as an intravenous infusion, over a minimum of 30 minutes 3 times every 4 weeks (3q4wk). Due to severe ocular toxicity, participants switched to receive Tisotumab vedotin at 2.0 mg/kg, administered as an intravenous infusion once every 3 weeks (1q3w).
- Part 2 Cohort Expansion: Cohort 5 1q3w Ovarian: Participants with the indication of ovarian cancer, received Tisotumab vedotin 2.0 mg/kg, administered as an intravenous infusion, over a minimum of 30 minutes, once every 3 weeks (1q3w); the revised dose and schedule due to severe ocular toxicity observed at 1.2 mg/kg 3q4wk.
- Part 2: Cohort Expansion: Cohort 6 1q3w Cervical: Participants with the indication of cervical cancer, received Tisotumab vedotin 2.0 mg/kg, administered as an intravenous infusion, over a minimum of 30 minutes, once every 3 weeks (1q3w); the revised dose and schedule due to severe ocular toxicity observed at 1.2 mg/kg 3q4wk.
Period: Part 1: Dose Level 1 (Weeks 1-16)
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2 Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2 Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Started | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1: Dose Level 2 (Week 17-48)
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2 Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2 Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Started | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Patient Choice | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Investigator Judgment | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Miscellaneous | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Cohort Expansion
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2 Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2 Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Started | 0 | 0 | 11 | 3 | 1 | 5 | 1 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not Completed | 0 | 0 | 11 | 3 | 1 | 4 | 1 | 3
Not completed — Patient Choice | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Disease Progression | 0 | 0 | 3 | 2 | 1 | 4 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 6 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical: Participants with the indication of ovarian cancer, received Tisotumab vedotin 1.2 mg/kg (the recommended dose for phase II trials [RP2D] from the Dose Escalation part), administered as an intravenous infusion, over a minimum of 30 minutes 3 times every 4 weeks (3q4wk).
- Total: Total of all reporting groups
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2 Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2 Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical | Total
Number analyzed (Participants) | 3 | 6 | 11 | 3 | 1 | 5 | 1 | 3 | 33
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 0 | 3 | 10 | 3 | 1 | 4 | 1 | 3 | 25
  From 65 to 84 years | 3 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 11 | 3 | 1 | 5 | 1 | 3 | 29
  Male | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 6 | 10 | 3 | 1 | 5 | 1 | 3 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 5 | 10 | 3 | 1 | 5 | 1 | 3 | 31
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 0 | 0 | 6 | 3 | 0 | 2 | 0 | 2 | 13
  United States | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 4
  Denmark | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 5
  United Kingdom | 1 | 1 | 4 | 0 | 1 | 2 | 1 | 1 | 11
Weight [Median (Full Range); unit: kg] — Population: The study was conducted in two parts; Part 1 Dose Escalation and Part 2 Cohort Expansion. Each part was analyzed separately.
  kg
    Part 1: Dose Escalation: number analyzed (Participants) | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 9
    Part 1: Dose Escalation | 80.0 [76.3 to 80.0] | 67.5 [48.1 to 85.0] |  |  |  |  |  |  | 74.7 [48.1 to 85.0]
    Part 2: Cohort Expansion: number analyzed (Participants) | 0 | 0 | 11 | 3 | 1 | 5 | 1 | 3 | 24
    Part 2: Cohort Expansion |  |  | 66.8 [40.0 to 89.6] | 55.2 [41.7 to 63.5] | 57.8 [57.8 to 57.8] | 72.0 [52.8 to 79.3] | 96.8 [96.8 to 96.8] | 65.3 [60.5 to 65.5] | 64.8 [40.0 to 96.8]
Height [Median (Full Range); unit: cm] — Population: The study was conducted in two parts; Part 1 Dose Escalation and Part 2 Cohort Expansion. Each part was analyzed separately.
  cm
    Part 1: Dose Escalation: number analyzed (Participants) | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 9
    Part 1: Dose Escalation | 171.0 [168.0 to 171.4] | 162.0 [156.0 to 175.0] |  |  |  |  |  |  | 168.0 [156.0 to 175.0]
    Part 2: Cohort Expansion: number analyzed (Participants) | 0 | 0 | 11 | 3 | 1 | 5 | 1 | 3 | 24
    Part 2: Cohort Expansion |  |  | 159.0 [154.0 to 174.0] | 157.0 [148.0 to 161.0] | 160.6 [160.6 to 160.6] | 168.0 [159.0 to 177.8] | 170.5 [170.5 to 170.5] | 161.0 [156.0 to 162.0] | 160.8 [148.0 to 177.8]
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] — Population: The study was conducted in two parts; Part 1 Dose Escalation and Part 2 Cohort Expansion. Each part was analyzed separately.
  kg/m^2
    Part 1: Dose Escalation: number analyzed (Participants) | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 9
    Part 1: Dose Escalation | 27.4 [26.0 to 28.3] | 25.5 [19.8 to 27.8] |  |  |  |  |  |  | 25.7 [19.8 to 28.3]
    Part 2: Cohort Expansion: number analyzed (Participants) | 0 | 0 | 11 | 3 | 1 | 5 | 1 | 3 | 24
    Part 2: Cohort Expansion |  |  | 26.4 [16.9 to 32.5] | 22.4 [16.1 to 29.0] | 22.4 [22.4 to 22.4] | 24.0 [18.7 to 28.5] | 33.3 [33.3 to 33.3] | 24.9 [23.3 to 26.9] | 25.1 [16.1 to 33.3]

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants Who Experience at Least One Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Baseline to end of follow-up; maximum time of follow-up was 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
Participants | 3 | 6

2. Primary Outcome: Part 2: Number of Participants Who Experience at Least One Adverse Event (AE)
Description: as for outcome 1
Time Frame: Baseline to end of trial (Part 2), up to 36 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian: Participants with the indication of ovarian cancer, received Tisotumab vedotin 1.2 mg/kg (RP2D from the Dose Escalation part), administered as an intravenous infusion, over a minimum of 30 minutes 3 times every 4 weeks (3q4wk). Due to severe ocular toxicity, participants switched to receive Tisotumab vedotin at 2.0 mg/kg, administered as an intravenous infusion once every 3 weeks (1q3w).
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2 Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 11 | 3 | 1 | 5 | 1 | 3
Participants | 11 | 3 | 1 | 5 | 0 | 3

3. Primary Outcome: Part 1: Number of Participants Who Experienced at Least One or More Serious Adverse Event (SAE)
Description: A SAE is defined as an AE that met one or more of the following criteria/outcomes which were classified as serious:
  Required inpatient hospitalization or prolongation of existing hospitalization. Resulted in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions.
  Was a congenital anomaly/birth defect. Medically important determined by the investigator. Resulted in death. Was life-threatening.
Time Frame: Baseline to end of follow-up; maximum time of follow-up was 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
Participants | 1 | 2

4. Primary Outcome: Part 2: Number of Participants Reporting One or More Serious Adverse Events (SAE)
Description: as for outcome 3
Time Frame: Baseline to end of trial (Part 2), up to 36 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian: Participants with the indication of ovarian cancer, received Tisotumab vedotin 2.0 mg/kg, administered as an intravenous infusion, over a minimum of 30 minutes, once every 3 weeks (1q3w); the revised dose and schedule due to severe ocular toxicity observed at 1.2 mg/kg 3q4wk.
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 11 | 3 | 1 | 5 | 1 | 3
Participants | 9 | 2 | 0 | 2 | 0 | 1

5. Primary Outcome: Part 1: Number of Participants Reporting One or More Infusion-related Adverse Events
Description: An infusion-related adverse event (AE) was defined as an AE occurring during infusion where the onset date and time of the event occurred within infusion time (+24 hours), and the event was judged as related to tisotumab vedotin by the investigator.
Time Frame: Day 1, Day 8 & Day 15 (+1 day) until end of treatment (Part 1), approximately 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
Participants | 2 | 4

6. Primary Outcome: Part 2: Number of Participants Reporting One or More Infusion-related Adverse Events
Description: as for outcome 5
Time Frame: Day 1, Day 8 & Day 15 (+1 day) until end of trial (Part 2), up to 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 11 | 3 | 1 | 5 | 1 | 3
Participants | 4 | 2 | 1 | 1 | 0 | 1

7. Primary Outcome: Part 1: Number of Participants Reporting One or More Common Terminology Criteria for Adverse Events (CTCAE) Grade >=3 Adverse Events
Description: A CTCAE AE was determined using the CTCAE grading systems based on NCI-CTCAE version 4.03 assessed by the investigator.
Time Frame: Baseline to end of follow-up; maximum time of follow-up was 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
Participants | 1 | 3

8. Primary Outcome: Part 2: Number of Participants Reporting One or More Common Terminology Criteria for Adverse Events (CTCAE) Grade >=3 Adverse Events
Description: A CTCAE AE was determined using the CTCAE grading systems based on NCI-CTCAE version 4.03 assessed by the investigator.
Time Frame: Baseline to end of trial (Part 2), up to 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 11 | 3 | 1 | 5 | 1 | 3
Participants | 10 | 2 | 0 | 3 | 0 | 1

9. Primary Outcome: Part 1: Number of Participants Reporting One or More Treatment-related Adverse Events
Description: A treatment-related AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; which has a causal relationship with the treatment.
Time Frame: Baseline to end of follow-up; maximum time of follow-up was 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
Participants | 3 | 6

10. Primary Outcome: Part 2: Number of Participants Reporting One or More Treatment-related Adverse Events
Description: as for outcome 9
Time Frame: Baseline to end of trial (Part 2), up to 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 11 | 3 | 1 | 5 | 1 | 3
Participants | 9 | 3 | 1 | 5 | 0 | 3

11. Secondary Outcome: Part 1: Number of Participants With Markedly Abnormal Laboratory Values
Description: The number of participants with any markedly abnormal standard safety laboratory values collected throughout study. Markedly abnormal laboratory values are defined as any grade >=3 laboratory abnormality events.
Time Frame: Baseline to end of follow-up; maximum time of follow-up was 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
Participants | 0 | 6

12. Secondary Outcome: Part 2: Number of Participants With Markedly Abnormal Laboratory Values
Description: as for outcome 11
Time Frame: Baseline to end of trial (Part 2), up to 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 11 | 3 | 1 | 5 | 1 | 3
Participants | 5 | 2 | 0 | 3 | 1 | 3

13. Secondary Outcome: Part 1: Number of Participants Who Experienced a Skin Rash
Time Frame: Baseline to end of follow-up; maximum time of follow-up was 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
Participants | 0 | 4

14. Secondary Outcome: Part 2: Number of Participants Who Experienced a Skin Rash
Time Frame: Baseline to end of trial (Part 2), up to 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 11 | 3 | 1 | 5 | 1 | 3
Participants | 2 | 0 | 1 | 1 | 0 | 1

15. Secondary Outcome: Part 1: Number of Participants Who Experienced a Bleeding Event
Time Frame: Baseline to end of trial (Part 1), up to 72 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
Participants | 3 | 5

16. Secondary Outcome: Part 2: Number of Participants Who Experienced a Bleeding Event
Time Frame: Baseline to end of trial (Part 2), up to 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 11 | 3 | 1 | 5 | 1 | 3
Participants | 7 | 3 | 1 | 5 | 0 | 2

17. Secondary Outcome: Part 1: Number of Participants Who Experienced a Neuropathy Event
Time Frame: Baseline to end of follow-up; maximum time of follow-up was 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
Participants | 1 | 3

18. Secondary Outcome: Part 2: Number of Participants Who Experienced a Neuropathy Event
Time Frame: Baseline to end of trial (Part 2), up to 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 11 | 3 | 1 | 5 | 1 | 3
Participants | 3 | 1 | 0 | 2 | 0 | 1

19. Secondary Outcome: Part 1: AUC0-t: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of Last Quantifiable Concentration for Tisotumab Vedotin (HuMax-TF-ADC)
Time Frame: Before infusion, end of infusion (+15 minutes), and +2 hours post infusion on days 1, 8 and 15, + 24 hours 1st infusion (Day 2), + 24 hours 3rd infusion (Day 16), + 72 hours 3rd infusion (Day 18), + 168 hours 3rd infusion (Day 22) of Cycle 1
Population: Insufficient samples were taken in Cycle 2 and beyond to calculate PK parameters, therefore only Cycle 1 is reported. Cycle 1 is an overall value, calculated over the entire cycle.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
h*µg/mL
  Cycle 1 | 3336 (7.3) | 5317 (34.6)
  Cycle 1 Day 1 | 867 (17.6) | 1328 (48.0)
  Cycle 1 Day 8 | 1603 (16.2) | 2216 (11.7)
  Cycle 1 Day 15 | 789 (15.6) | 1411 (94.2)

20. Secondary Outcome: Part 2: AUC0-t: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of Last Quantifiable Concentration for Tisotumab Vedotin (HuMax-TF-ADC)
Description: Due to severe ocular toxicity, participants switched to receive Tisotumab vedotin at 2.0 mg/kg administered as an intravenous infusion, over a minimum of 30 minutes, once every 3 weeks (1q3wk). Data has only been provided for participants who received the original dosing schedule of 3 times every 4 weeks (3q4wk).
Time Frame: Before infusion, end of infusion (+15 minutes) and +2 hours post infusion on day 1, and before infusion on days 8 and 15 of Cycle 1
Population: Insufficient samples were collected for cohorts 3-6 to calculate PK parameters. Insufficient samples were taken in Cycle 2 and beyond to calculate PK parameters, only Cycle 1 is reported. Cycle 1 is an overall value, calculated over the cycle. Includes data for all randomized participants for whom data were available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 11 | 3 | 0 | 0 | 0 | 0
h*µg/mL
  Cycle 1 | 2267 (24.8) | 1755 (19.1) |  |  |  |
  Cycle 1 Dose 1 | 1889 (29.3) | 1412 (11.9) |  |  |  |
  Cycle 1 Dose 2: number analyzed (Participants) | 9 | 3 | 0 | 0 | 0 | 0
  Cycle 1 Dose 2 | 150 (56.2) | 123 (85.4) |  |  |  |
  Cycle 1 Dose 3: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0 | 0
  Cycle 1 Dose 3 | 410 (26.4) | 204 (71.3) |  |  |  |

21. Secondary Outcome: Part 1: AUCinf: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Tisotumab Vedotin (HuMax-TF-ADC)
Description: Data is only available for Part 1, for Part 2 inadequate samples were collected after the third dose to define a terminal phase.
Time Frame: Before infusion, end of infusion (+15 minutes), and +2 hours post infusion on days 1, 8 and 15, + 24 hours 1st infusion (Day 2), +24 hours 3rd infusion (Day 16), +72 hours 3rd infusion (Day 18), +168 hours 3rd infusion (Day 22) of Cycle 1
Population: Insufficient samples were taken in Cycle 2 and beyond to calculate PK parameters, therefore only Cycle 1 is reported. Includes data for all randomized participants for whom data were available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 2 | 4
h*µg/mL | 920 (3.6) | 1106 (21.3)

22. Secondary Outcome: Part 1: Cmax: Maximum Observed Plasma Concentration for Tisotumab Vedotin (HuMax-TF-ADC)
Time Frame: Before infusion, end of infusion (+15 minutes), and +2 hours post infusion on days 1, 8, and 15, +24 hours 1st infusion (Day 2), +24 hours 3rd infusion (Day 16), +72 hours 3rd infusion (Day 18), and +168 hours 3rd infusion (Day 22) of Cycle 1
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
µg/mL
  Cycle 1 | 21.2 (14.5) | 30.7 (10.1)
  Cycle 1 Day 1 | 20.2 (17.9) | 28.7 (12.1)
  Cycle 1 Day 8 | 20.9 (14.1) | 28.0 (8.9)
  Cycle 1 Day 15 | 19.9 (11.8) | 26.8 (21.6)

23. Secondary Outcome: Part 2: Cmax: Maximum Observed Plasma Concentration for Tisotumab Vedotin (HuMax-TF-ADC)
Description: as for outcome 20
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 11 | 3 | 0 | 0 | 0 | 0
µg/mL
  Cycle 1 | 28.2 (34.5) | 19.5 (17.6) |  |  |  |
  Cycle 1 Dose 1 | 28.2 (34.5) | 19.5 (17.6) |  |  |  |
  Cycle 1 Dose 2: number analyzed (Participants) | 9 | 3 | 0 | 0 | 0 | 0
  Cycle 1 Dose 2 | 1.00 (42.0) | 1.13 (112.2) |  |  |  |
  Cycle 1 Dose 3: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0 | 0
  Cycle 1 Dose 3 | 3.85 (24.5) | 1.85 (77.6) |  |  |  |

24. Secondary Outcome: Part 1: Tmax: Time to Reach the Maximum Plasma Concentration for Tisotumab Vedotin (HuMax-TF-ADC)
Time Frame: as for outcome 22
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
hours
  Cycle 1 | 5.864 (172.022) | 5.061 (166.177)
  Cycle 1 Day 1 | 0.747 (11.547) | 0.873 (79.228)
  Cycle 1 Day 8 | 0.717 (0.000) | 0.846 (86.481)
  Cycle 1 Day 15 | 1.141 (81.075) | 1.084 (73.110)

25. Secondary Outcome: Part 2: Tmax: Time to Reach the Maximum Plasma Concentration for Tisotumab Vedotin (HuMax-TF-ADC)
Description: as for outcome 20
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 11 | 3 | 0 | 0 | 0 | 0
hours
  Cycle 1 | 0.75 (68.49) | 0.58 (22.85) |  |  |  |
  Cycle 1 Dose 1 | 0.75 (68.49) | 0.58 (22.85) |  |  |  |
  Cycle 1 Dose 2: number analyzed (Participants) | 9 | 3 | 0 | 0 | 0 | 0
  Cycle 1 Dose 2 | 165.06 (75.01) | 106.93 (55.38) |  |  |  |
  Cycle 1 Dose 3: number analyzed (Participants) | 6 | 3 | 0 | 0 | 0 | 0
  Cycle 1 Dose 3 | 71.23 (24.35) | 80.37 (20.24) |  |  |  |

26. Secondary Outcome: Part 1: Trough Concentration (Ctrough) Steady State Plasma Pharmacokinetic for Tisotumab Vedotin (HuMax-TF-ADC)
Description: Data is only available for Part 1, for Part 2 inadequate samples were collected to fully evaluate separate PK parameters after doses 1, 2, and 3.
Time Frame: Before infusion of Day 1, 8 and 15 of Cycle 1
Population: Insufficient samples were taken in Cycle 2 and beyond to calculate PK parameters, therefore only Cycle 1 is reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
ng/mL
  Cycle 1 Day 1 | 30.0 (0) | 30.0 (0)
  Cycle 1 Day 8 | 797.3 (22.1) | 1328.5 (191.8)
  Cycle 1 Day 15 | 912.1 (23.7) | 989.0 (44.3)

27. Secondary Outcome: Part 1: Terminal Phase Elimination Half-life (T1/2) for Tisotumab Vedotin (HuMax-TF-ADC)
Description: Data is only available for Part 1, for Part 2 inadequate samples were collected after the third dose to define a terminal phase, and therefore t1/2 could not be determined.
Time Frame: as for outcome 22
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Groups:
- Part 1: Dose Escalation: Cohort 1 3q4wk 0.9mg/kg: Tisotumab vedotin 0.9 mg/kg was administered as an intravenous infusion, over a minimum of 30 minutes, 3 times every 4 weeks (3q4wk).
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 4
hours | 40.45 (24.78) | 48.15 (16.47)

28. Secondary Outcome: Part 1: Total Clearance (CL) of Tisotumab Vedotin (HuMax-TF-ADC)
Description: Data is only available for Part 1, for Part 2 inadequate pharmacokinetic samples were collected after the third dose to define a terminal phase, and therefore CL could not be determined.
Time Frame: as for outcome 22
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h/kg
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 2 | 4
mL/h/kg | 0.979 (3.561) | 1.085 (21.476)

29. Secondary Outcome: Part 1: Apparent Volume of Distribution (Vz) for Tisotumab Vedotin (HuMax-TF-ADC)
Description: Data is only available for Part 1, for Part 2 inadequate samples were collected after the third dose to define a terminal phase, and therefore Vz could not be determined.
Time Frame: as for outcome 22
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/kg
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 2 | 4
mL/kg | 66.75 (6.67) | 75.37 (14.89)

30. Secondary Outcome: Part 1: AUC0-t: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of Last Quantifiable Concentration for Total HuMax-TF (Conjugated and Non-conjugated)
Time Frame: as for outcome 22
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
h*µg/mL
  Cycle 1 | 3916 (7.3) | 5573 (15.0)
  Cycle 1 Day 1 | 1058 (15.0) | 1530 (34.7)
  Cycle 1 Day 8 | 1750 (16.2) | 2460 (8.5)
  Cycle 1 Day 15 | 1012 (25.7) | 1426 (28.6)

31. Secondary Outcome: Part 2: AUC0-t: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of Last Quantifiable Concentration for Total HuMax-TF (Conjugated and Non-conjugated)
Description: as for outcome 20
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 11 | 3 | 0 | 0 | 0 | 0
h*µg/mL
  Cycle 1 | 2660 (20.0) | 1948 (35.2) |  |  |  |
  Cycle 1 Dose 1 | 1980 (24.5) | 460 (84.5) |  |  |  |
  Cycle 1 Dose 2: number analyzed (Participants) | 9 | 3 | 0 | 0 | 0 | 0
  Cycle 1 Dose 2 | 299 (55.0) | 192 (80.9) |  |  |  |
  Cycle 1 Dose 3: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0 | 0
  Cycle 1 Dose 3 | 679 (25.7) | 291 (89.9) |  |  |  |

32. Secondary Outcome: Part 1: AUCinf: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Total HuMax-TF (Conjugated and Non-conjugated)
Description: as for outcome 21
Time Frame: as for outcome 22
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 2 | 6
h*µg/mL | 1268 (14.4) | 1594 (24.6)

33. Secondary Outcome: Part 1: Cmax: Maximum Observed Plasma Concentration for Total HuMax-TF (Conjugated and Non-conjugated)
Time Frame: as for outcome 22
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
µg/mL
  Cycle 1 | 22.1 (9.1) | 31.7 (11.9)
  Cycle 1 Day 1 | 20.3 (14.3) | 30.2 (34.7)
  Cycle 1 Day 8 | 21.0 (6.3) | 29.2 (6.6)
  Cycle 1 Day 15 | 20.9 (12.0) | 29.2 (16.2)

34. Secondary Outcome: Part 2: Cmax: Maximum Observed Plasma Concentration for Total HuMax-TF (Conjugated and Non-conjugated)
Description: as for outcome 20
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 11 | 3 | 0 | 0 | 0 | 0
µg/mL
  Cycle 1 | 27.5 (36.4) | 20.6 (18.6) |  |  |  |
  Cycle 1 Dose 1 | 27.5 (36.4) | 20.6 (18.6) |  |  |  |
  Cycle 1 Dose 2: number analyzed (Participants) | 9 | 3 | 0 | 0 | 0 | 0
  Cycle 1 Dose 2 | 2.00 (41.6) | 1.91 (105.0) |  |  |  |
  Cycle 1 Dose 3: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0 | 0
  Cycle 1 Dose 3 | 6.39 (24.6) | 3.68 (66.1) |  |  |  |

35. Secondary Outcome: Part 1: Tmax: Time to Reach the Maximum Plasma Concentration for Total HuMax-TF (Conjugated and Non-conjugated)
Time Frame: as for outcome 22
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
hours
  Cycle 1 | 36.445 (99.474) | 14.003 (117.534)
  Cycle 1 Day 1 | 0.747 (11.547) | 0.893 (66.752)
  Cycle 1 Day 8 | 0.717 (0) | 0.869 (78.568)
  Cycle 1 Day 15 | 0.727 (4.784) | 0.896 (78.665)

36. Secondary Outcome: Part 2: Tmax: Time to Reach the Maximum Plasma Concentration for Total HuMax-TF (Conjugated and Non-conjugated)
Description: as for outcome 20
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 11 | 3 | 0 | 0 | 0 | 0
hours
  Cycle 1 | 0.86 (73.61) | 0.58 (22.85) |  |  |  |
  Cycle 1 Dose 1 | 0.86 (73.61) | 0.58 (22.85) |  |  |  |
  Cycle 1 Dose 2: number analyzed (Participants) | 9 | 3 | 0 | 0 | 0 | 0
  Cycle 1 Dose 2 | 165.06 (75.01) | 106 (55.38) |  |  |  |
  Cycle 1 Dose 3: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0 | 0
  Cycle 1 Dose 3 | 71.23 (24.35) | 80.37 (20.24) |  |  |  |

37. Secondary Outcome: Part 1: Terminal Phase Elimination Half-life (T1/2) for Total HuMax-TF (Conjugated and Non-conjugated)
Description: as for outcome 27
Time Frame: as for outcome 22
Population: Insufficient samples were taken in Cycle 2 and beyond to calculate PK parameters, therefore only Cycle 1 is reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
hours | 49.56 (17.35) | 49.34 (19.18)

38. Secondary Outcome: Part 1 and Part 2: Total Clearance (CL) of Total HuMax-TF (Conjugated and Non-conjugated)
Description: CL could not be estimated for Part 1 or Part 2 participants due to insufficient number of samples taken.
Time Frame: 0 to 2 hours post-dose on days 1, 8, 15, +24 hrs 1st infusion, +24 hrs 3rd infusion, +72 hrs 3rd infusion, +168 hrs 3rd infusion (Part 1) and 0 to 2 hours post-dose on day 1, and pre-dose days 8 and 15 (Part 2) of Cycle 1
Population: CL could not be estimated for Part 1 or Part 2 participants.
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

39. Secondary Outcome: Part 1 & Part 2: Apparent Volume of Distribution (Vz) for Total HuMax-TF (Conjugated and Non-conjugated)
Description: Vz could not be estimated for Part 1 or Part 2 participants due to insufficient number of samples taken.
Time Frame: as for outcome 38
Population: Vz could not be estimated for Part 1 or Part 2 participants.
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

40. Secondary Outcome: Part 1: Trough Concentration (Ctrough) Steady State Plasma Pharmacokinetic for Total HuMax-TF (Conjugated and Non-conjugated)
Description: Data is only available for Part 1, for Part 2, inadequate samples were collected to fully evaluate separate PK parameters after doses 1, 2, and 3.
Time Frame: Before infusion on Day 1, 8 and 15 of Cycle 1
Population: Insufficient samples were taken in Cycle 2 and beyond to calculate PK parameters, therefore only Cycle 1 is reported. Data includes all randomized participants for whom data were available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 2 | 6
  Cycle 1 Day 1 | 150.0 (0.0) | 150.0 (0.0)
  Cycle 1 Day 8 | 1273.1 (23.4) | 1252.2 (53.3)
  Cycle 1 Day 15 | 1625.1 (24.4) | 1863.8 (46.6)

41. Secondary Outcome: Part 1: AUC0-t: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of Last Quantifiable Concentration for Free Toxin (MMAE)
Time Frame: as for outcome 22
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
h*ng/mL
  Cycle 1 | 885 (27.1) | 968 (59.7)
  Cycle 1 Day 1 | 185 (48.1) | 185 (75.3)
  Cycle 1 Day 8 | 180 (14.1) | 236 (75.5)
  Cycle 1 Day 15 | 506 (25.3) | 520 (51.3)

42. Secondary Outcome: Part 2: AUC0-t: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of Last Quantifiable Concentration for Free Toxin (MMAE)
Description: as for outcome 20
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 11 | 3 | 0 | 0 | 0 | 0
h*ng/mL
  Cycle 1 | 920 (74.5) | 1049 (89.4) |  |  |  |
  Cycle 1 Dose 1 | 439 (69.3) | 393 (100.0) |  |  |  |
  Cycle 1 Dose 2: number analyzed (Participants) | 9 | 3 | 0 | 0 | 0 | 0
  Cycle 1 Dose 2 | 378 (121.3) | 366 (77.9) |  |  |  |
  Cycle 1 Dose 3: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0 | 0
  Cycle 1 Dose 3 | 713 (49.9) | 494 (121.7) |  |  |  |

43. Secondary Outcome: Part 1: Cmax: Maximum Observed Plasma Concentration for Free Toxin (MMAE)
Time Frame: as for outcome 22
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
ng/mL
  Cycle 1 | 2.76 (23.7) | 2.88 (52.4)
  Cycle 1 Day 1 | 1.46 (54.7) | 1.38 (78.4)
  Cycle 1 Day 8 | 1.18 (19.8) | 1.54 (75.4)
  Cycle 1 Day 15 | 2.76 (23.7) | 2.88 (52.4)

44. Secondary Outcome: Part 2: Cmax: Maximum Observed Plasma Concentration for Free Toxin (MMAE)
Description: as for outcome 20
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 11 | 3 | 0 | 0 | 0 | 0
ng/mL
  Cycle 1 | 3.9 (97.0) | 3.6 (101.4) |  |  |  |
  Cycle 1 Dose 1 | 1.9 (110.5) | 1.5 (80.4) |  |  |  |
  Cycle 1 Dose 2: number analyzed (Participants) | 9 | 3 | 0 | 0 | 0 | 0
  Cycle 1 Dose 2 | 2.47 (136.4) | 2.50 (81.1) |  |  |  |
  Cycle 1 Dose 3: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0 | 0
  Cycle 1 Dose 3 | 3.78 (81.6) | 3.23 (125.0) |  |  |  |

45. Secondary Outcome: Part 1: Tmax: Time to Reach the Maximum Plasma Concentration for Free Toxin (MMAE)
Time Frame: as for outcome 22
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
hours
  Cycle 1 | 392.024 (3.256) | 373.366 (6.290)
  Cycle 1 Day 1 | 44.568 (114.567) | 32.001 (125.788)
  Cycle 1 Day 8 | 10.354 (165.509) | 20.837 (106.094)
  Cycle 1 Day 15 | 54.511 (20.424) | 32.537 (63.879)

46. Secondary Outcome: Part 2: Tmax: Time to Reach the Maximum Plasma Concentration for Free Toxin (MMAE)
Description: as for outcome 20
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 11 | 3 | 0 | 0 | 0 | 0
hours
  Cycle 1 | 307.05 (36.52) | 410.61 (3.82) |  |  |  |
  Cycle 1 Dose 1 | 160.56 (5.66) | 162.19 (1.71) |  |  |  |
  Cycle 1 Dose 2: number analyzed (Participants) | 9 | 3 | 0 | 0 | 0 | 0
  Cycle 1 Dose 2 | 164.82 (56.71) | 106.93 (55.38) |  |  |  |
  Cycle 1 Dose 3: number analyzed (Participants) | 6 | 2 | 0 | 0 | 0 | 0
  Cycle 1 Dose 3 | 78.37 (50.26) | 80.37 (20.24) |  |  |  |

47. Secondary Outcome: Part 1: Trough Concentration (Ctrough) Steady State Plasma Pharmacokinetic for Free Toxin (MMAE)
Description: as for outcome 26
Time Frame: Before infusion on Day 1, 8 and 15 of Cycle 1
Population: Insufficient samples were taken in Cycle 2 and beyond to calculate PK parameters, therefore only Cycle 1 is reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
pg/mL
  Cycle 1 Day 1 | 12.50 (0) | 12.50 (0)
  Cycle 1 Day 8 | 853.42 (22.93) | 1061.28 (87.81)
  Cycle 1 Day 15 | 1013.22 (14.47) | 1384.29 (83.43)

48. Secondary Outcome: Part 1: Number of Participants With a Positive Anti-drug Antibody (ADA) Immunogenicity Result
Time Frame: Baseline to end of follow-up; maximum follow-up was 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
Participants | 0 | 0

49. Secondary Outcome: Part 2: Number of Participants With a Positive Anti-drug Antibody (ADA) Immunogenicity Result
Time Frame: Baseline to end of trial (Part 2), up to 36 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian: Participants with the indication of ovarian cancer, received Tisotumab vedotin 2.0 mg/kg, administered as an intravenous infusion, over a minimum of 30 minutes, once every 3 weeks (1q3w); the revised dose and schedule due to severe ocular toxicity.
- Part 2: Cohort Expansion: Cohort 6 1q3w Cervical: Participants with the indication of cervical cancer, received Tisotumab vedotin 2.0 mg/kg, administered as an intravenous infusion, over a minimum of 30 minutes, once every 3 weeks (1q3w); the revised dose and schedule due to severe ocular toxicity.
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 11 | 3 | 1 | 5 | 1 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0

50. Secondary Outcome: Part 1: Number of Patients Who Experienced Anti-tumor Activity Measured by Tumor Shrinkage
Time Frame: Baseline to end of trial (Part 1), up to 72 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
Participants | 1 | 3

51. Secondary Outcome: Part 2: Anti-tumor Activity Measured by Percentage of Change in Sum of Lesion Measurements
Time Frame: Baseline to end of trial (Part 2), up to 36 weeks
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 11 | 3 | 1 | 5 | 1 | 3
percentage of change | -17.34 (43.388) | 32.78 (83.933) | -63.27 (NA) — Only 1 participant is included in this arm, therefore Standard deviation cannot be calculated. | 0.74 (21.877) | 0 (NA) — Only 1 participant is included in this arm, therefore Standard deviation cannot be calculated. | 11.76 (27.658)

52. Secondary Outcome: Part 1: Response Evaluation Based on PSA (Prostate Specific Antigen [Prostate Cancer]): Percentage Change From Baseline to End of Study
Time Frame: Baseline to end of follow-up; maximum follow-up was 24 weeks
Population: PSA is only assessed for participants with prostate cancer. 2 participants in Part 1 Cohort 1 and 1 participant in Part 1 Cohort 2 had the indication of prostate cancer.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 2 | 1
percentage of change | 23.42 (61.686) | 12.97 (NA) — Only 1 participant is included in the analysis, therefore Standard deviation cannot be calculated.

53. Secondary Outcome: Part 1: Response Evaluation Based on CA125 (Cancer Antigen 125 [Ovarian and Endometrial Cancer]): Percentage of Change From Baseline to End of Study
Time Frame: Baseline to end of follow-up; maximum follow-up was 24 weeks
Population: CA 125 is only assessed for participants with ovarian and endometrial cancer, 1 participant in Cohort 1 and 1 participant in Cohort 2 had the indication of ovarian or endometrial cancer. No participants from Cohort 1 with the indication of ovarian and endometrial Cancer had results at the End of Study visit.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 0 | 1
percentage of change |  | 186.21 (NA) — Only 1 participant was included in the analysis, therefore Standard deviation could not calculated.

54. Secondary Outcome: Part 2: Response Evaluation Based on CA125 (Cancer Antigen 125 [Ovarian and Endometrial Cancer]): Percentage of Change From Baseline to End of Study
Time Frame: Baseline to end of trial (Part 2), up to 36 week
Population: CA 125 was only assessed for participants with Ovarian cancer. No participants from Cohort 5 participated in the End of Trial visit.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian
Number analyzed (Participants) | 8 | 1 | 0
percentage of change | -31.75 (36.235) | -32.50 (NA) — Only 1 participant was included in the analysis, therefore Standard deviation could not be calculated. |

55. Secondary Outcome: Part 1: Best Overall Response (OR)
Description: Best OR (by investigators assessment) was the best response recorded from the start of the treatment until disease progression or death. Complete response: the disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm. Based on non-target lesions, complete response was defined as disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (< 10 mm short axis).
  Partial response (PR): ≥ 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum of LDs.
  Stable disease: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum of LDs while in trial. Based on non-target lesions, stable disease was defined as persistence of 1 or more non-target lesion(s) or/and maintenance of tumor marker level above the normal limits.
Time Frame: Baseline to end of trial (Part 1), up to 72 weeks
Measure: Number; unit: participants
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
participants
  Complete Response | 0 | 0
  Partial Response | 0 | 1
  Stable Disease | 2 | 3
  Progressive Disease | 1 | 1
  Not Evaluable | 0 | 1

56. Secondary Outcome: Part 2: Best Overall Response (OR)
Description: as for outcome 55
Time Frame: Baseline to end of trial (Part 2), up to 36 weeks
Measure: Number; unit: participants
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 11 | 3 | 1 | 5 | 1 | 3
participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 3 | 1 | 1 | 2 | 0 | 0
  Stable Disease | 3 | 0 | 0 | 2 | 0 | 2
  Progressive Disease | 2 | 2 | 0 | 1 | 1 | 1
  Not Evaluable | 3 | 0 | 0 | 0 | 0 | 0

57. Secondary Outcome: Part 1: Number of Participants Who Experienced Disease Control
Description: Participants were defined as having disease control at a specific time point if they had an evaluation of complete response (CR) or partial response (PR) at the time point (with a window of +/- 7 days) or had an evaluation of stable disease (SD), PR or CR at any point from the time point minus 7 days or later.
Time Frame: 6, 12, 24 and 36 weeks post first infusion (Part 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 3 | 6
Participants
  6 Weeks: Disease Control - Yes | 2 | 3
  6 Weeks: Disease Control - No | 1 | 3
  12 Weeks: Disease Control - Yes | 0 | 0
  12 Weeks: Disease Control - No | 3 | 6
  24 Weeks: Disease Control - Yes | 0 | 0
  24 Weeks: Disease Control - No | 3 | 6
  36 Weeks: Disease Control - Yes | 0 | 0
  36 Weeks: Disease Control - No | 3 | 6

58. Secondary Outcome: Part 2: Number of Participants Who Experienced Disease Control
Description: as for outcome 57
Time Frame: 6, 12, 24 and 36 weeks post first infusion (Part 2)
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 11 | 3 | 1 | 5 | 1 | 3
Participants
  6 Weeks: Disease Control - Yes | 6 | 1 | 1 | 4 | 0 | 2
  6 Weeks: Disease Control - No | 5 | 2 | 0 | 1 | 1 | 1
  12 Weeks: Disease Control - Yes | 2 | 1 | 1 | 2 | 0 | 1
  12 Weeks: Disease Control - No | 9 | 2 | 0 | 3 | 1 | 2
  24 Weeks: Disease Control - Yes | 0 | 0 | 0 | 1 | 0 | 0
  24 Weeks: Disease Control - No | 11 | 3 | 1 | 4 | 1 | 3
  36 Weeks: Disease Control - Yes | 0 | 0 | 0 | 0 | 0 | 0
  36 Weeks: Disease Control - No | 11 | 3 | 1 | 5 | 1 | 3

59. Secondary Outcome: Part 1: Progression Free Survival (PFS)
Description: Progression-free survival was defined as the time in weeks from date of first dose until the date of disease progression or death, whichever is earliest.
Time Frame: Baseline to end of follow-up; maximum time of follow-up was 24 weeks
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 2 | 1
weeks | 11.3 [7.3 to 15.3] | NA [7.1 to NA] — Could not be estimated due to the low number of events disease progression or death.

60. Secondary Outcome: Part 2: Progression Free Survival (PFS)
Description: as for outcome 59
Time Frame: Baseline to end of trial (Part 2), up to 36 weeks
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 4 | 2 | 1 | 4 | 1 | 3
weeks | 10.7 [2.0 to NA] — Could not be estimated due to the low number of events disease progression or death. | 8.0 [4.3 to NA] — Could not be estimated due to the low number of events disease progression or death. | 22.0 [NA to NA] — Could not be estimated due to the low number of events disease progression or death. | 14.0 [9.1 to NA] — Could not be estimated due to the low number of events disease progression or death. | 5.0 [NA to NA] — Could not be estimated due to the low number of events disease progression or death. | 11.9 [11.0 to 17.1]

61. Secondary Outcome: Part 1: Duration of Response
Description: Duration of response was defined as as the number of days from the first documentation of objective tumor response (complete response [CR] or partial response [PR]) to the date of first progressive disease (PD) or death.
Time Frame: Baseline to end of trial (Part 1), up to 72 weeks
Population: Duration of Response could not be estimated in the Dose Escalation or the Cohort Expansion parts of the trial because patients with a confirmed response were discontinued due to toxicity or other reason different from progressive disease (PD) or death.
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg
Number analyzed (Participants) | 0 | 0

62. Secondary Outcome: Part 2: Duration of Response
Description: as for outcome 61
Time Frame: Baseline to end of trial (Part 2), up to 36 weeks
Population: as for outcome 61
Arm/Group | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2: Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2: Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Part 1: Dose Escalation: Baseline to follow-up; maximum time of follow-up was 24 weeks. Part 2: Cohort Expansion: Baseline to a maximum of 36 weeks.
Groups:
- Part 2 Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian: Participants with the indication of ovarian cancer, received Tisotumab vedotin 1.2 mg/kg (RP2D from the Dose Escalation part), administered as an intravenous infusion, over a minimum of 30 minutes 3 times every 4 weeks (3q4wk). Due to severe ocular toxicity, participants switched to receive Tisotumab vedotin at 2.0 mg/kg, administered as an intravenous infusion, once every 3 weeks (1q3w).
- Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical: Participants with the indication of cervical cancer, received Tisotumab vedotin 1.2 mg/kg (RP2D from the Dose Escalation part), administered as an intravenous infusion, over a minimum of 30 minutes 3 times every 4 weeks (3q4wk). Due to severe ocular toxicity, participants switched to receive Tisotumab vedotin at 2.0 mg/kg, administered as an intravenous infusion, once every 3 weeks (1q3w).
Arm/Group | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical | Part 2 Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical | Part 2 Cohort Expansion: Cohort 5 1q3w Ovarian | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 1/11 | 0/3 | 0/1 | 0/5 | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/6 | 9/11 | 2/3 | 0/1 | 2/5 | 0/1 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 10/11 | 3/3 | 1/1 | 5/5 | 0/1 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg (N=3) | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg (N=6) | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian (N=11) | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical (N=3) | Part 2 Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian (N=1) | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical (N=5) | Part 2 Cohort Expansion: Cohort 5 1q3w Ovarian (N=1) | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical (N=3)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Symblepharon (Eye disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Dose Escalation: Cohort 1 3q4wk 0.9 mg/kg (N=3) | Part 1: Dose Escalation: Cohort 2 3q4wk 1.2 mg/kg (N=6) | Part 2: Cohort Expansion: Cohort 1 3q4wk Ovarian (N=11) | Part 2: Cohort Expansion: Cohort 2 3q4wk Cervical (N=3) | Part 2 Cohort Expansion: Cohort 3 3q4wk - 1q3w Ovarian (N=1) | Part 2: Cohort Expansion: Cohort 4 3q4wk - 1q3w Cervical (N=5) | Part 2 Cohort Expansion: Cohort 5 1q3w Ovarian (N=1) | Part 2: Cohort Expansion: Cohort 6 1q3w Cervical (N=3)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (5) | 5 (5) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 5 (6) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 4 (4) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 3 (4) | 1 (1) | 0 (0) | 4 (6) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue blistering (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (6) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal discharge (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 2 (2) | 6 (7) | 5 (6) | 0 (0) | 0 (0) | 3 (8) | 0 (0) | 1 (1)
Escherichia vaginitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 5 (5) | 7 (8) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 2 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (9) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2) | 6 (8) | 1 (1) | 1 (1) | 4 (6) | 0 (0) | 2 (3)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 3 (4) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cell death (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 5 (5) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Symblepharon (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meibomianitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Punctate keratitis (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Episcleritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Keratopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vital dye staining cornea present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine output increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (4) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiation proctitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 12 months but less than 18 months from the end of study (database lock). The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT02552121/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/21/NCT02552121/SAP_001.pdf